CLINICAL TRIAL: NCT01765439
Title: The Effect of VSL#3 (Original De Simone Formulation) Probiotic Preparation on the Bile Acid Metabolism in Patients With Inflammatory Bowel Disease
Brief Title: The Effect of VSL#3 Probiotic Preparation on the Bile Acid Metabolism in Patients With Inflammatory Bowel Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Iscare i.v.f., Czech Republic (Unknown); CD Investments srl (Unknown); University Of Perugia (Other); University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Martin Lenicek, assistant professor, Charles University, Czech Republic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VSL#3-2013-CR
Record Dates: First submitted 2013-01-07; First posted 2013-01-10 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Crohn Disease; Ulcerative Colitis
Keywords: bile acids; metabolism; probiotics
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CD resected (Experimental): Patients with Crohn´s disease with the history of single resection (<60 cm) of distal leum.
  Interventions: Dietary Supplement: VSL#3 (Original De Simone formulation)
- UC unoperated (Experimental): Patients with ulcerative colitis without history of gut resection.
  Interventions: Dietary Supplement: VSL#3 (Original De Simone formulation)
- UC IPAA (Experimental): Patients with ulcerative colitis after proctocolectomy and ileal pouch-anal anastomosis(IPAA).
  Interventions: Dietary Supplement: VSL#3 (Original De Simone formulation)
- Healthy volunteers (Experimental): Subjects without any sign of disease of the digestive tract.
  Interventions: Dietary Supplement: VSL#3 (Original De Simone formulation)

INTERVENTIONS:
Dietary Supplement: VSL#3 (Original De Simone formulation) — Study subjects will receive two sachets of VSL#3 probiotic (ie 2x900 billions of live bacteria) per day (one in the morning, one in the evening). The intervention period will be 6 weeks (plus or minus 5 days).

SUMMARY:
The aim of the study is to determine, whether administration of VSL#3 (Original De Simone formulation) probiotic preparation can alter the bile acid metabolism in patients with inflammatory bowel disease.

DETAILED DESCRIPTION:
VSL#3 (Original De Simone formulation, further abbreviated as VSL#3), a potent probiotic preparation, has been tested as an adjuvant therapy in inflammatory bowel diseases (IBD), chronic unspecific inflammatory disorders of the gastrointestinal tract (the most frequent forms of IBD are Crohn's disease (CD) and ulcerative colitis (UC)). VSL#3 has been shown to improve symptoms of IBD both in animal models and in humans-the most impressive results have been observed in preventing of pouchitis in UC patients. Several possible mechanisms of its action have been suggested, including change in gut microbial diversity, immunomodulatory function (upregulation of interleukine-10), etc., however, the list is probably far from complete.

Bile acids (BA) play an important role in the gastrointestinal tract - besides facilitating fat (and protein) digestion and resorption, they act as general antimicrobial agents within the small intestine (maintaining the small intestine more or less microbe-free), colonic microflora modifiers, intestinal innate immunity regulators, and importantly as signalling molecules on the liver-intestine/intestine-liver axis. Under pathological conditions (such as BA malabsorption) BA can worsen the IBD symptoms (namely diarrhoea), by irritating colonic mucosa or by inducing colonic secretion of electrolytes.

The study hypothesis is that the beneficial effect of VSL#3 might be partially explained by alteration of BA metabolism. There exists a complex crosstalk between gut microflora and BA: BA affect microbial growth, whereas BA structure is modified by bacteria (deconjugation, 7 α dehydroxylation). Several observations might support this hypothesis: VSL#3 ameliorates symptoms of radiation or chemotherapy induced diarrhoea, as well as diarrhoea of critically ill patients - conditions, that can be caused by BA malabsorption. Similarly, oxalate absorption (closely related to BA malabsorption) has been shown to be lowered by VSL#3. The main question to be addressed in the proposed study is, therefore, whether VSL#3 administration can somehow change metabolism of bile acids (BA).

Additionally, urinary metabolite levels are strongly influenced by differences in the intestinal microbiota, since both gut bacterial metabolism, and shared metabolism by the host and bacterial species ('co-metabolism'), generate specific metabolic products. Such metabolites may therefore be used as markers of microbial metabolic activity, reflecting systemic, functional differences. This application of urinary metabolic profiling avoids the technical difficulties, and methodological differences, found in molecular studies of the intestinal microbiota in IBD, which have contributed to often discrepant findings. Specific urinary metabolites related to gut microbial metabolism differ between CD patients, UC patients, and controls. The emerging technique of urinary NMR-based metabolic profiling with multivariate analysis was able to distinguish these cohorts. This study should address the question, whether VSL#3 administration changes the nuclear magnetic resonance-based urinary metabolomic profile.

ELIGIBILITY:
Inclusion Criteria:

Arm CD resected

* confirmed diagnosis of Crohn´s disease (at least 6 months)
* history of single resection of terminal ileum (at least 6 months before inclusion)
* maximum length of resected ileum is 60 cm
* no signs of disease activity (clinical, endoscopical, laboratory)
* stable medication

Arm UC unoperated

* confirmed diagnosis of ulcerative colitis (at least 6 months)
* no signs of disease activity (clinical, endoscopical, laboratory)
* stable medication

Arm UC IPAA

* confirmed diagnosis of ulcerative colitis (at least 6 months)
* proctocolectomy and IPAA (at least 3 months before inclusion)
* no signs of disease activity (clinical, endoscopical, laboratory)
* stable medication

Arm Healthy volunteers

* no signs of gastrointestinal disorder
* initial laboratory examination within normal range (blood count, liver function tests, C-reactive protein, Fe, ferritin, fecal calprotectin)

Exclusion Criteria:

* use of bile acids
* use of bile acids sequestrants
* use of farnesoid X receptor agonists/antagonists
* recent colonoscopy(less than 1 month before inclusion)
* diabetes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-02; Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Alteration in the rate of bile acid synthesis | Baseline and 6 weeks (plus or minus 5 days)
  Will be assessed as difference between serum levels of fibroblast growth factor 19 and C4 at baseline and 6 weeks, respectively.

SECONDARY OUTCOMES:
Change of the spectrum of bile acids in stools and plasma | Baseline and 6 weeks (plus or minus 5 days).
Change of a metabolomic profile in urine | Baseline and 6 weeks (plus or minus 5 days).

OTHER OUTCOMES:
Change of the disease activity | Baseline and 6 weeks (plus or minus 5 days).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lenicek, MD, Ph.D., Principal Investigator — Charles University, Czech Republic
Locations (1):
- Iscare I.V.F., Prague, Czechia